CLINICAL TRIAL: NCT01623596
Title: A 12-month, Prospective, Randomized, Active-controlled, Open-label Study to Evaluate the Patient Retention of Fingolimod vs. Approved First-line Disease Modifying Therapies in Adults With Relapsing Remitting Multiple Sclerosis (PREFERMS)
Brief Title: Evaluation of Patient Retention of Fingolimod vs. Currently Approved Disease Modifying Therapy in Patients With Relapsing Remitting Multiple Sclerosis.
Acronym: PREFERMS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CFTY720DUS09
Record Dates: First submitted 2012-06-18; First posted 2012-06-20 (Estimated); Results first posted 2018-01-12 (Actual); Last update posted 2021-01-05 (Actual); Status verified 2019-03

CONDITIONS: Relapsing Remitting Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting | interventions — Fingolimod Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fingolimod (Experimental)
  Interventions: Drug: Fingolimod
- Disease Modifying Therapy (Active Comparator): 2 classes - Interferon Beta preparation (Exctavia, Betaseron, Rebif, Avonex) or glatiramer acetate (Copaxone)
  Interventions: Drug: Disease Modifying therapy

INTERVENTIONS:
Drug: Fingolimod
  Arms: Fingolimod
Drug: Disease Modifying therapy
  Arms: Disease Modifying Therapy

SUMMARY:
A 12 month study where 852 patients with relapsing remitting MS will be randomized 1:1 to fingolimod or approved disease modifying therapy. Patients will be be treatment naive or have only been treated with one class of DMT (Interferon beta preparation or glatiramer acetate) . Patients will be able to switch to different treatment for safety, efficacy, tolerability or convenience during the study.

Primary objective is to evaluate efficacy of fingolimod by assessing patients retention on treatment. Secondary objectives are to compare reasons for discontinuation, adverse events, cognitive impairment, medication satisfaction and change in brain volume measured by MRI.

DETAILED DESCRIPTION:
852 Patients with relapsing remitting MS will be randomized 1:1 to fingolimod or approved first line DMTs. Patients must be either treatment naive or have received treatment with only one class of treatment (interferon beta preparation or glatiramer acetate) . Patients previously treated with DMT and randomized to the DMT arm may not remain on the same treatment for the study and will have to switch to a different class (i.e., previously treated with glatiramer acetate will switch to interferon beta preparaption, previously treated with interferon beta preparation will swtich to glatiramer acetate).

Entry criteria at screening include but are not limited to, age 18-65, diagnosis with RRMS, EDSS < or equal to 6, not pregnant or planning pregnancy and women of childbearing potential willing to use contraception throughout the study.

Exclusion criteria include but are not limited to - prior exposure to fingolimod, history of malignancy within 5 years, other than RRMS types of MS, other diseases of the immune system, active macular edema, systemic bacterial, viral or fungal infections, patients without vaccine against varicella zoster, receipt of live or attentuated vaccines within a month of screening, history of various cardiac conditions, presence of certain ECG abnormalities, resting heart rate < 45 bpm, symptomatic bradycardia, recurrent syncope, severe untreated sleep apnea, severe pulmonary conditions, various hepatic conditions, certain neurologic disorders, pregnancy.

Patients may switch treatment before 3 months for safety reasons only, after 3 months for safety, efficacy, tolerability or convenience. Treatment switch during the study may be to any of study approved treatments irrespective of prior treatment.

Patients randomized to fingolimod will need to have 6 hours of observation for signs and symptoms of bradycardia following administration of the first dose. Extended observation or overnight observation may be necessary under certain circumstances. Primary objective is to evaluate efficacy of fingolimod by assessing patients retention on treatment. Secondary objectives are to compare reasons for discontinuation, adverse events, cognitive impairment, medication satisfaction and change in brain volume measured by MRI. Exploratory objectives include annualized relapse rate, OCT, MRI evaluations, biomarkers and patient reported outcome measures.

ELIGIBILITY:
Inclusion Criteria:

1. written informed consent must be obtained prior to any assessment being performed.
2. Male and female patients aged 18-65 years inclusive.
3. Patients diagnosed with relapsing remitting MS, defined by the 2010 revised McDonald criteria (Pollman et al, 2011) (Appendix 1).
4. EDSS score of less than or equal to 6.
5. Patients naive to treatment or who have been treated with no more than one class of DMT previously (interferon β preparation or glatiramer acetate), and who, per investigator judgment, may benefit from a change of treatment class.
6. Patients who have been treated with DMF for less than 2 months total exposure and who have a normal lymphocyte count at screening.
7. Women of childbearing potential must have a negative urine and serum β-human chorionic gonadotropin (β-hCG) pregnancy test at screening and at baseline.
8. Before entry women must be:

   * Post menopausal for at least 1 year, or
   * Surgically sterile (have had a hysterectomy or bilateral oophorectomy, tubal ligation or otherwise incapable of pregnancy, or
   * Practicing a highly effective method of birth control if sexually active, including hormonal prescription oral contraceptives, contraceptive injections, contraceptive patch, intrauterine device, double barrier method (e.g., condoms, diaphragm or cervical cap with spermicidal foam, cream or gel), or male partner sterilization consistent with local regulations regarding use of birth control methods for patients participating in clinical trials, for the duration of their participation in the study, or
   * Not heterosexually active (patients who are not heterosexually active at screening must agree to utilize a highly effective method of birth control if they become heterosexually active during their participation in the study) 4.2 Exclusion criteria

<!-- -->

1. Use of other investigational drugs within 30 days of screening.
2. History of hypersensitivity to any of the study drugs or to drugs of similar chemical classes.
3. Prior exposure to fingolimod or any other S1P receptor modulating compounds.
4. History or presence of malignancy of any organ system (other than successfully treated basal or squamous cell carcinoma of the skin or stage 0 carcinoma of the cervix), treated or untreated, within the past 5 years, regardless of whether there is evidence of local recurrence or metastases.
5. Patients diagnosed with Secondary Progressive Multiple Sclerosis (SPMS) or Primary Progressive MS (PPMS).
6. Patients with a history of chronic disease of the immune system other than MS or a known immunodeficiency syndrome.
7. Patients who have been treated with:

   • Natalizumab, mitoxantrone, cladribine, rituximab, alemtuzumab, ofatumumab, ocrelizumab at any time before randomization

   • Immunoglobulins, or pulse of corticosteroids with more than 6 months cumulative exposure

   • Immunosuppressive/chemotherapeutic medications (e.g., methotrexate, azathioprine, cyclophosphamide, cellcept, Cytoxan, IVIG) with more than 6 months of cumulative exposure and within 6 months prior to randomization

   • Corticosteroids or adrenocorticotropic hormones in the past 30 days before randomization. Patients that require corticosteroids for a relapse during the screening period may be rescreened 30 days after the last dose.
8. History of treatment with both classes of approved first line DMT (interferon β preparation and glatiramer acetate) or DMF exposure of 2 months or longer.
9. Patients with uncontrolled diabetes mellitus (HbA1c > 7%).
10. Diagnosis of macular edema during the screening phase. Patients with a history of macular edema will be allowed to enter the study provided that they do not have macular edema at the screening visit.
11. Patients with active systemic bacterial, viral or fungal infections, or known to have AIDS, Hepatitis B, Hepatitis C infection or positive HIV antibody, Hepatitis B surface antigen or Hepatitis C antibody tests.
12. Patients without history of chickenpox or without vaccination against varicella-zoster virus at screening (patients may be vaccinated and rescreened one month or longer after vaccination).
13. Patients who have received any live or live attenuated vaccines (including for varicella-zoster or measles) within 1 month prior to baseline.
14. Patients with any medically unstable condition as assessed by the investigator.
15. Patients with a history of the following cardiovascular conditions:

    • Cardiac arrest.

    • myocardial infarction, unstable angina, stroke, transient ischemic attack, decompensated heart failure requiring hospitalization, or Class III/IV heart failure (Appendix 3).

    • Congestive heart failure.

    • Hypertension that is not controlled with prescribed medications. These patients may be rescreened if blood pressure is stabilized with treatment.

    • Cerebrovascular disease.

    • History or presence of Mobitz Type II 2nd degree or 3rd degree AV block or sick sinus syndrome, unless patient has a pacemaker.

    • Patients at higher risk of symptomatic bradycardia or heart block because of a coexisting medical condition or certain concomitant medications.

    • Patients randomized to the fingolimod arm with prolonged QTc interval at screening (corrected QT interval > 450 ms in males and > 470 ms in females); for patients randomized to the fingolimod treatment arm before dosing (baseline) or during the 6-hour observation period; and those patients at additional risk for QT prolongation (e.g., hypokalemia, hypomagnesemia, congenital long-QT syndrome), or on a concomitant therapy with QT prolonging drugs with a known risk of Torsades de pointes (e.g., citalopram, chlorpromazine, haloperidol, methadone, erythromycin).
    * Patients receiving class Ia or Class III antiarrhythmic drugs (Appendix 6)
    * Patients receiving concurrent therapy with drugs that slow the heart rate or atrioventricular conduction (e.g., beta blockers, digoxin, or heart-rate slowing calcium channel blockers such as diltiazem, verapamil or digoxin). The possibility to switch to drugs that do not slow the heart rate or atrioventricular conduction should be evaluated by the physician prescribing these drugs before initiating fingolimod treatment.
    * History of sick sinus syndrome or sinoatrial heart block.
    * Resting heart rate of < 45 bpm or symptomatic bradycardia
    * Recurrent syncope
    * Severe untreated sleep apnea
16. Patients with severe pulmonary conditions (including severe respiratory disease, pulmonary fibrosis, active tuberculosis, severe or poorly controlled asthma).
17. Patients with any of the following hepatic conditions:

    • Chronic liver or biliary disease
    * Total bilirubin greater than upper limit of normal (ULN) at screening unless in the context of Gilbert's syndrome
    * Conjugated bilirubin greater than the ULN at screening
    * AST (SGOT), ALT (SGPT) greater than 3 times ULN at screening
    * Alkaline phosphatase (AP) greater than 1.5 times the ULN at screening
18. Serum creatinine greater than 2.0 mg/dL (176.5 µmol/L) at screening.
19. Patients with the following neurological/psychiatric disorders:

    * History of substance abuse (drug or alcohol) in the past five years as determined by the investigator
    * Progressive neurological disorder other than MS which may affect study participation as determined by the investigator
    * Any serious psychiatric condition that may interfere with the patient's ability to cooperate and comply with the study procedures as determined by the investigator
20. Women who are pregnant or nursing (lactating) or planning to become pregnant.
21. Any condition that in the opinion of the investigator, would compromise the well-being of the patient or the conduct of the study, or prevent the patient from meeting or performing study requirements.
22. Pre-planned surgery or medical procedure that would interfere with the conduct of the study.
23. Employee of the sponsor, investigator or study center, with direct involvement in the proposed study or other studies under the direction of that investigator or study center, as well as family members of the employees or the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 881 (Actual)
Dates: Start 2012-06-08 (Actual); Primary Completion 2015-07-13 (Actual); Study Completion 2015-07-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (115):
- United States (114):
  - Novartis Investigative Site, Cullman, Alabama
  - Novartis Investigative Site, Phoenix, Arizona
  - Novartis Investigative Site, Sun City, Arizona
  - Novartis Investigative Site, Tucson, Arizona
  - Novartis Investigative Site, Sherwood, Arkansas
  - Novartis Investigative Site, Fullerton, California
  - Novartis Investigative Site, Oceanside, California
  - Novartis Investigative Site, San Francisco, California
  - Novartis Investigative Site, Walnut Creek, California
  - Novartis Investigative Site, Basalt, Colorado
  - Novartis Investigative Site, Boulder, Colorado
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Fort Collins, Colorado
  - Novartis Investigative Site, Fairfield, Connecticut
  - Novartis Investigative Site, New London, Connecticut
  - Novartis Investigative Site, Dover, Delaware
  - Novartis Investigative Site, Atlantis, Florida
  - Novartis Investigative Site, Bradenton, Florida
  - Novartis Investigative Site, Delray Beach, Florida
  - Novartis Investigative Site, Hollywood, Florida
  - Novartis Investigative Site, Jacksonville, Florida
  - Novartis Investigative Site, North Palm Beach, Florida
  - Novartis Investigative Site, Plantation, Florida
  - Novartis Investigative Site, Pompano Beach, Florida
  - Novartis Investigative Site, Port Charlotte, Florida
  - Novartis Investigative Site, Port Orange, Florida
  - Novartis Investigative Site, Sarasota, Florida
  - Novartis Investigative Site, St. Petersburg, Florida
  - Novartis Investigative Site, Tallahassee, Florida
  - Novartis Investigative Site, Tampa, Florida
  - Novartis Investigative Site, West Palm Beach, Florida
  - Novartis Investigative Site, Atlanta, Georgia
  - Novartis Investigative Site, Columbus, Georgia
  - Novartis Investigative Site, Decatur, Georgia
  - Novartis Investigative Site, Suwanee, Georgia
  - Novartis Investigative Site, Flossmoor, Illinois
  - Novartis Investigative Site, Northbrook, Illinois
  - Novartis Investigative Site, Anderson, Indiana
  - Novartis Investigative Site, Indianapolis, Indiana
  - Novartis Investigative Site, Des Moines, Iowa
  - Novartis Investigative Site, Overland Park, Kansas
  - Novartis Investigative Site, Wichita, Kansas
  - Novartis Investigative Site, Hawesville, Kentucky
  - Novartis Investigative Site, Lexington, Kentucky
  - Novartis Investigative Site, Madisonville, Kentucky
  - Novartis Investigative Site, Alexandria, Louisiana
  - Novartis Investigative Site, Baton Rouge, Louisiana
  - Novartis Investigative Site, New Orleans, Louisiana
  - Novartis Investigative Site, Annapolis, Maryland
  - Novartis Investigative Site, Fulton, Maryland
  - Novartis Investigative Site, New Bedford, Massachusetts
  - Novartis Investigative Site, North Dartmouth, Massachusetts
  - Novartis Investigative Site, Springfield, Massachusetts
  - Novartis Investigative Site, Watertown, Massachusetts
  - Novartis Investigative Site, Worcester, Massachusetts
  - Novartis Investigative Site, Kalamazoo, Michigan
  - Novartis Investigative Site, Traverse City, Michigan
  - Novartis Investigative Site, Nixa, Missouri
  - Novartis Investigative Site, North Kansas City, Missouri
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Las Vegas, Nevada
  - Novartis Investigative Site, Flemington, New Jersey
  - Novartis Investigative Site, Teaneck, New Jersey
  - Novartis Investigative Site, Toms River, New Jersey
  - Novartis Investigative Site, Albuquerque, New Mexico
  - Novartis Investigative Site, Albany, New York
  - Novartis Investigative Site, Amherst, New York
  - Novartis Investigative Site, Kingston, New York
  - Novartis Investigative Site, Latham, New York
  - Novartis Investigative Site, New York, New York
  - Novartis Investigative Site, Patchogue, New York
  - Novartis Investigative Site, The Bronx, New York
  - Novartis Investigative Site, Asheville, North Carolina
  - Novartis Investigative Site, Charlotte, North Carolina
  - Novartis Investigative Site, Greensboro, North Carolina
  - Novartis Investigative Site, Greenville, North Carolina
  - Novartis Investigative Site, Raleigh, North Carolina
  - Novartis Investigative Site, Salisbury, North Carolina
  - Novartis Investigative Site, Winston-Salem, North Carolina
  - Novartis Investigative Site, Grand Forks, North Dakota
  - Novartis Investigative Site, Akron, Ohio
  - Novartis Investigative Site, Bellevue, Ohio
  - Novartis Investigative Site, Canton, Ohio
  - Novartis Investigative Site, Cincinnati, Ohio
  - Novartis Investigative Site, Columbus, Ohio
  - Novartis Investigative Site, Dayton, Ohio
  - Novartis Investigative Site, Toledo, Ohio
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Eugene, Oregon
  - Novartis Investigative Site, Greensburg, Pennsylvania
  - Novartis Investigative Site, Hershey, Pennsylvania
  - Novartis Investigative Site, Pittsburgh, Pennsylvania
  - Novartis Investigative Site, Cranston, Rhode Island
  - Novartis Investigative Site, Old Point Station, South Carolina
  - Novartis Investigative Site, Spartanburg, South Carolina
  - Novartis Investigative Site, Cordova, Tennessee
  - Novartis Investigative Site, Knoxville, Tennessee
  - Novartis Investigative Site, Nashville, Tennessee
  - Novartis Investigative Site, Colleyville, Texas
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, Lubbock, Texas
  - Novartis Investigative Site, North Richland Hills, Texas
  - Novartis Investigative Site, Plano, Texas
  - Novartis Investigative Site, Round Rock, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Orem, Utah
  - Novartis Investigative Site, Alexandria, Virginia
  - Novartis Investigative Site, Norfolk, Virginia
  - Novartis Investigative Site, Vienna, Virginia
  - Novartis Investigative Site, Bothell, Washington
  - Novartis Investigative Site, Seattle, Washington
  - Novartis Investigative Site, Tacoma, Washington
  - Novartis Investigative Site, Morgantown, West Virginia
  - Novartis Investigative Site, Neenah, Wisconsin
- Novartis Investigative Site, Guaynabo, Puerto Rico

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=34

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 62 Fingolimod arm participants discontinued: 57 discontinued before treatment switch, and 5 discontinued after treatment switch
  100 MS-DMT arm participants discontinued before treatment switch: 57 discontinued before treatment switch, and 43 discontinued after treatment switch
Pre-assignment Details: Patient disposition was summarized on the Randomized Set.
  Randomized Set (RS): consists of all participants who were assigned randomization numbers.
Groups:
- Fingolimod: fingolimod 0.5 mg once a day
Period: Overall Study
Arm/Group | Fingolimod | Disease Modifying Therapy
Started | 436 | 439
On Randomized Treatment | 352 | 125
On Switched Treatment | 22 | 214
Completed | 374 | 339
Not Completed | 62 | 100
Not completed — Abnormal laboratory values | 2 | 0
Not completed — Administrative problems | 9 | 13
Not completed — Adverse Event | 20 | 29
Not completed — Death | 0 | 2
Not completed — Lost to Follow-up | 12 | 16
Not completed — Withdrawal by Subject | 13 | 31
Not completed — Patient no longer requires study drug | 1 | 0
Not completed — Protocol Violation | 0 | 6
Not completed — Lack of Efficacy | 5 | 3

BASELINE CHARACTERISTICS:
Population: Randomized set (RS): consists of all patients who were assigned randomization numbers. The participants in this set were called randomized participants. This set was used to summarize participant disposition, demographic and baseline characteristics, and protocol deviation information. Participants were grouped according to randomized treatment.
Groups:
- Disease Modifying Therapy (MS_DMT): 2 classes - Interferon Beta preparation (Exctavia, Betaseron, Rebif, Avonex) or glatiramer acetate (Copaxone)
- Total: Total of all reporting groups
Arm/Group | Fingolimod | Disease Modifying Therapy (MS_DMT) | Total
Number analyzed (Participants) | 436 | 439 | 875
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.5 (10.84) | 41.9 (10.39) | 41.7 (10.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 311 | 329 | 640
  Male | 125 | 110 | 235

OUTCOME MEASURES:

1. Primary Outcome: Participant Retention Rate Over 12 Months
Description: Comparison effectiveness of fingolimod versus approved first-line disease modifying therapies by measuring the rate of participant retention on randomized treatment over a 12-month period (Full analysis set)
Time Frame: at 12 months
Population: Full analysis set includes all the patients who received at least one dose of study medication and had information on the primary end point.
Measure: Number; unit: participants
Groups:
- Disease Modifying Therapy (MS-DMT): 2 classes - Interferon Beta preparation (Exctavia, Betaseron, Rebif, Avonex) or glatiramer acetate (Copaxone)
Arm/Group | Fingolimod | Disease Modifying Therapy (MS-DMT)
Number analyzed (Participants) | 436 | 439
participants | 352 | 125

2. Secondary Outcome: Primary and Secondary Reasons for Discontinuation From Randomized Treatment: Randomized Set
Description: Reasons for discontinuation in participants treated with fingolimod vs. DMT over 12 months of treatment
  Total discontinued (Primary reason): Fingolimod arm: 27, MS-DMT arm: 27 = 54 participants
  Total discontinued (Secondary reason): Fingolimod arm: 257, MS-DMT arm: 256 = 513 participants
  Throughout the study, investigators evaluated each patient for occurrence of randomized treatment discontinuation and determined the primary and secondary reasons for such discontinuation. At every visit, the investigator evaluated the patients and determined if they should continue on randomized treatment or change to alternative treatment. Treatment discontinuation was a clinically meaningful measure related to safety, efficacy, and tolerability over time, reflecting the therapeutic effectiveness of study treatment.
Time Frame: at 12 months
Population: Randomized set (RS): consists of all patients who were assigned randomization numbers.
  The patients in this set were called randomized patients. This set was used to summarize patient disposition, demographic and baseline characteristics, and protocol deviation information. Patients were grouped according to randomized treatment.
Measure: Number; unit: participants
Arm/Group | Fingolimod | Disease Modifying Therapy (MS-DMT)
Number analyzed (Participants) | 436 | 439
participants
  Occurrence of relapse (Primary reason) | 5 | 14
  Disease activity present in MRI (Primary reason) | 0 | 6
  Injection site reaction (Primary reason) | 0 | 61
  Flu-like symptoms (Primary reason) | 0 | 34
  Lipoatrophy (Primary reason) | 0 | 1
  Depression (Primary reason) | 1 | 4
  Hepatic side effects (Primary reason) | 7 | 3
  Spasticity (Primary reason) | 0 | 1
  Infection (Primary reason) | 0 | 0
  Macular edema (Primary reason) | 1 | 0
  Bradycardia (Primary reason) | 0 | 0
  Needle phobia (Primary reason) | 0 | 13
  Inconvenient administration (Primary reason) | 0 | 33
  Frequency of injections (Primary reason) | 0 | 29
  Neutralizing antibodies present (Primary reason) | 0 | 0
  Other (Primary reason) | 13 | 58
  Occurrence of relapse (Secondary reason) | 0 | 3
  Disease activity present in MRI (Secondary reason) | 2 | 5
  Injection site reaction (Secondary reason) | 0 | 40
  Flu-like symptoms (Secondary reason) | 1 | 16
  Lipoatrophy (Secondary reason) | 0 | 1
  Depression (Secondary reason) | 0 | 6
  Hepatic side effects (Secondary reason) | 5 | 0
  Spasticity (Secondary reason) | 1 | 2
  Infection (Secondary reason) | 0 | 0
  Macular edema (Secondary reason) | 1 | 0
  Bradycardia (Secondary reason) | 0 | 0
  Needle phobia (Secondary reason) | 0 | 18
  Inconvenient administration (Secondary reason) | 0 | 55
  Frequency of injections (Secondary reason) | 0 | 45
  Neutralizing antibodies present (Secondary reason) | 0 | 0
  Other (Secondary reason) | 17 | 65

3. Secondary Outcome: Change From Baseline of Symbol Digit Modalities Test (SDMT) Scores (Oral Test) by Visit (Randomized Treatment / Randomized Phase)
Description: Summary statistics Compare cognitive impairment measured by Symbol Digit Modalities Test (SDMT) scores. The SDMT score and its change from baseline value were summarized by visit. For the change from baseline values at each visit, ANCOVA adjusted for treatment naivety, corresponding baseline values, and age was performed for treatment comparisons
  The SDMT measures the time to pair abstract symbols with specific numbers. The test requires elements of attention, visuoperceptual processing, working memory, and psychomotor speed. The score is the number of correctly coded items from 0-110 in 90 seconds. The total score provides a measure of the speed and accuracy of symbol-digit substitution.
  NOTE: Higher scores indicate better performance.
Time Frame: baseline, 6 months, 12 months, and Last assessment which is either at Month 12 or at early discontinuation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SDMT score
Arm/Group | Fingolimod | Disease Modifying Therapy (MS-DMT)
Number analyzed (Participants) | 433 | 428
SDMT score
  Baseline (n=76,70): number analyzed (Participants) | 76 | 70
  Baseline (n=76,70) | 52.00 (12.12) | 51.60 (13.40)
  Change at 6 months (n=70,64): number analyzed (Participants) | 70 | 64
  Change at 6 months (n=70,64) | 2.20 (8.09) | 0.20 (10.13)
  Change at 12 months (n=58, 18): number analyzed (Participants) | 58 | 18
  Change at 12 months (n=58, 18) | 3.20 (7.09) | 1.40 (8.33)
  Change at Last assessment (n=73, 65): number analyzed (Participants) | 73 | 65
  Change at Last assessment (n=73, 65) | 3.30 (7.77) | 0.40 (9.47)

4. Secondary Outcome: Change From Baseline of Symbol Digit Modalities Test (SDMT) Scores (Written Test) by Visit (Randomized Treatment / Randomized Phase)
Description: as for outcome 3
Time Frame: baseline, 6 months, 12 months, Last assessment which is either at Month 12 or at early discontinuation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: SDMT score
Arm/Group | Fingolimod | Disease Modifying Therapy (MS-DMT)
Number analyzed (Participants) | 433 | 428
SDMT score
  Baseline (n=355,348): number analyzed (Participants) | 355 | 348
  Baseline (n=355,348) | 48.90 (18.26) | 48.50 (20.19)
  Change at 6 months (n=339,322): number analyzed (Participants) | 339 | 322
  Change at 6 months (n=339,322) | -0.50 (14.04) | 0.70 (13.16)
  Change at 12 months (n=282,105): number analyzed (Participants) | 282 | 105
  Change at 12 months (n=282,105) | 0.70 (16.02) | 0.40 (14.90)
  Change at Last assessment (n=342, 324): number analyzed (Participants) | 342 | 324
  Change at Last assessment (n=342, 324) | 0.80 (16.27) | 0.70 (13.95)

5. Secondary Outcome: Percent Change From Baseline in Brain Volume From Month 12 to Last Visit (Randomized)
Description: Summary statistics for percent change from month 12 in brain volume by visit (Randomized treatment / randomized phase) in patients treated with fingolimod vs.DMTs as measured by MRI
Time Frame: 12 months, and Last assessment which is either at Month 12 or at early discontinuation
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent change in brain volume
Arm/Group | Fingolimod | Disease Modifying Therapy
Number analyzed (Participants) | 433 | 428
percent change in brain volume
  Percent change at 12 months (n=323, 111): number analyzed (Participants) | 323 | 111
  Percent change at 12 months (n=323, 111) | -0.396 (0.7825) | -0.555 (0.7181)
  Percent change at Last assessment (n=370, 246): number analyzed (Participants) | 370 | 246
  Percent change at Last assessment (n=370, 246) | -0.385 (0.7690) | -0.420 (0.6423)

6. Secondary Outcome: Number of Satisfied Participants Per Medication Satisfaction Questionnaire (MSQ) Score
Description: Summary statistics for Medication Satisfaction Questionnaire[Question: "Overall, how satisfied are you with your current medication?"] (Randomized treatment / randomized phase): Fingolimod vs MS-DMT
Time Frame: Baseline, 1 month, 3 months, 6 months, 9 months, at 12 months & Last assessment during randomized phase which is either at Month 12 or at early discontinuation
Population: Full analysis set (FAS) includes all the patients who received at least one dose of study medication and had information on the primary end point.
Measure: Number; unit: participants
Groups:
- Disease Modifying Therapy (DS-DMT): 2 classes - Interferon Beta preparation (Exctavia, Betaseron, Rebif, Avonex) or glatiramer acetate (Copaxone)
Arm/Group | Fingolimod | Disease Modifying Therapy (DS-DMT)
Number analyzed (Participants) | 433 | 428
participants
  Baseline, Extremely dissatisfied | 10 (4.7) | 16 (7.2)
  Baseline, Very dissatisfied | 22 (10.3) | 13 (5.8)
  Baseline, Somewhat dissatisfied | 29 (13.6) | 39 (17.5)
  Baseline, Neither dissatisfied nor satisfied | 62 (29.0) | 61 (27.4)
  Baseline, Somewhat satisfied | 35 (16.4) | 46 (20.6)
  Baseline, Very satisfied | 42 (19.6) | 31 (13.9)
  Baseline, Extremely satisfied | 14 (6.5) | 17 (7.6)
  Baseline, Missing | 219 (0) | 205 (0)
  1 month, Extremely dissatisfied | 8 (1.9) | 29 (6.9)
  1 month, Very dissatisfied | 14 (3.3) | 37 (8.9)
  1 month, Somewhat dissatisfied | 8 (1.9) | 52 (12.4)
  1 month, Neither dissatisfied nor satisfied | 32 (7.5) | 74 (17.7)
  1 month, Somewhat satisfied | 52 (12.1) | 89 (21.3)
  1 month, Very satisfied | 161 (37.5) | 97 (23.2)
  1 month, Extremely satisfied | 154 (35.9) | 40 (9.6)
  1 month, Missing | 4 (0) | 10 (0)
  3 months, Extremely dissatisfied | 5 (1.2) | 19 (5.5)
  3 months, Very dissatisfied | 11 (2.7) | 38 (11.0)
  3 months, Somewhat dissatisfied | 11 (2.7) | 42 (12.1)
  3 months, Neither dissatisfied nor satisfied | 46 (11.1) | 53 (15.3)
  3 months, Somewhat satisfied | 43 (10.4) | 73 (21.1)
  3 months, Very satisfied | 153 (37.0) | 91 (26.3)
  3 months, Extremely satisfied | 144 (34.9) | 30 (8.7)
  3 months, Missing | 20 (0) | 82 (0)
  6 months, Extremely dissatisfied | 8 (2.0) | 9 (4.6)
  6 months, Very dissatisfied | 15 (3.8) | 11 (5.6)
  6 months, Somewhat dissatisfied | 11 (2.8) | 13 (6.6)
  6 months, Neither dissatisfied nor satisfied | 25 (6.3) | 24 (12.2)
  6 months, Somewhat satisfied | 57 (14.4) | 46 (23.5)
  6 months, Very satisfied | 130 (32.7) | 67 (34.2)
  6 months, Extremely satisfied | 151 (38.0) | 26 (13.3)
  6 months, Missing | 36 (0) | 232 (0)
  9 months, Extremely dissatisfied | 7 (1.9) | 4 (2.6)
  9 months, Very dissatisfied | 8 (2.2) | 6 (3.9)
  9 months, Somewhat dissatisfied | 12 (3.2) | 12 (7.8)
  9 months, Neither dissatisfied nor satisfied | 21 (5.7) | 15 (9.8)
  9 months, Somewhat satisfied | 42 (11.4) | 29 (19.0)
  9 months, Very satisfied | 135 (36.5) | 58 (37.9)
  9 months, Extremely satisfied | 145 (39.2) | 29 (19.0)
  9 months, Missing | 63 (0) | 275 (0)
  12 months, Extremely dissatisfied | 7 (2.0) | 3 (2.4)
  12 months, Very dissatisfied | 7 (2.0) | 4 (3.1)
  12 months, Somewhat dissatisfied | 11 (3.1) | 4 (3.1)
  12 months, Neither dissatisfied nor satisfied | 27 (7.7) | 8 (6.3)
  12 months, Somewhat satisfied | 34 (9.7) | 22 (7.3)
  12 months, Very satisfied | 115 (32.8) | 60 (47.2)
  12 months, Extremely satisfied | 150 (42.7) | 26 (20.5)
  12 months, Missing | 82 (0) | 301 (0)
  Last assessment, Extremely dissatisfied | 14 (3.3) | 46 (10.9)
  Last assessment, Very dissatisfied | 15 (3.5) | 61 (14.5)
  Last assessment, Somewhat dissatisfied | 23 (5.3) | 57 (13.5)
  Last assessment,Neither dissatisfied nor satisfied | 45 (10.5) | 58 (13.7)
  Last assessment, Somewhat satisfied | 43 (10.0) | 69 (16.4)
  Last assessment, Very satisfied | 128 (29.8) | 94 (22.3)
  Last assessment, Extremely satisfied | 162 (37.7) | 37 (8.8)
  Last assessment, Missing | 3 (0) | 6 (0)

ADVERSE EVENTS:
Groups:
- Fingolimod: Fingolimod
- MS DMT: MS DMT
Arm/Group | Fingolimod | MS DMT
Serious Adverse Events (participants affected / at risk) | 29/433 | 15/428
Other Adverse Events (participants affected / at risk) | 282/433 | 291/428
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod (N=433) | MS DMT (N=428)
Leukocytosis (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Bradycardia (Cardiac disorders) | 1 | 0
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Myocardial infarction (Cardiac disorders) | 1 | 0
Macular oedema (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 | 0
Gastric ulcer (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Jejunal ulcer (Gastrointestinal disorders) | 1 | 0
Pneumoperitoneum (Gastrointestinal disorders) | 1 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 1
Asthenia (General disorders) | 1 | 0
Localised oedema (General disorders) | 1 | 0
Systemic inflammatory response syndrome (General disorders) | 1 | 0
Biliary colic (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 0 | 1
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Bacteraemia (Infections and infestations) | 1 | 0
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 0
Pneumonia (Infections and infestations) | 2 | 0
Pneumonia influenzal (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 1 | 0
Tooth abscess (Infections and infestations) | 1 | 0
Viral infection (Infections and infestations) | 1 | 0
Gastrointestinal stoma complication (Injury, poisoning and procedural complications) | 1 | 0
Intentional overdose (Injury, poisoning and procedural complications) | 0 | 1
Pubis fracture (Injury, poisoning and procedural complications) | 1 | 0
Seroma (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Suture related complication (Injury, poisoning and procedural complications) | 1 | 0
Dehydration (Metabolism and nutrition disorders) | 2 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Mental impairment (Nervous system disorders) | 0 | 1
Multiple sclerosis relapse (Nervous system disorders) | 5 | 5
Optic neuritis (Nervous system disorders) | 1 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Sciatica (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 1 | 0
Agoraphobia (Psychiatric disorders) | 0 | 1
Anxiety (Psychiatric disorders) | 1 | 2
Depression (Psychiatric disorders) | 1 | 0
Homicidal ideation (Psychiatric disorders) | 1 | 0
Major depression (Psychiatric disorders) | 1 | 0
Panic disorder (Psychiatric disorders) | 0 | 1
Personality disorder (Psychiatric disorders) | 0 | 1
Suicidal ideation (Psychiatric disorders) | 2 | 0
Calculus urinary (Renal and urinary disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Abortion induced (Surgical and medical procedures) | 1 | 1
Haematoma (Vascular disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fingolimod (N=433) | MS DMT (N=428)
Lymphopenia (Blood and lymphatic system disorders) | 30 | 1
Diarrhoea (Gastrointestinal disorders) | 26 | 5
Nausea (Gastrointestinal disorders) | 29 | 22
Fatigue (General disorders) | 49 | 33
Influenza like illness (General disorders) | 12 | 64
Injection site erythema (General disorders) | 0 | 42
Injection site pain (General disorders) | 0 | 62
Injection site pruritus (General disorders) | 0 | 30
Injection site reaction (General disorders) | 0 | 50
Nasopharyngitis (Infections and infestations) | 41 | 22
Sinusitis (Infections and infestations) | 28 | 21
Upper respiratory tract infection (Infections and infestations) | 27 | 21
Urinary tract infection (Infections and infestations) | 23 | 16
Lymphocyte count decreased (Investigations) | 23 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 30 | 17
Back pain (Musculoskeletal and connective tissue disorders) | 29 | 14
Pain in extremity (Musculoskeletal and connective tissue disorders) | 18 | 23
Dizziness (Nervous system disorders) | 31 | 12
Headache (Nervous system disorders) | 40 | 41
Hypoaesthesia (Nervous system disorders) | 23 | 15
Migraine (Nervous system disorders) | 22 | 14
Paraesthesia (Nervous system disorders) | 22 | 17
Anxiety (Psychiatric disorders) | 13 | 24
Depression (Psychiatric disorders) | 26 | 29
Cough (Respiratory, thoracic and mediastinal disorders) | 25 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial